CLINICAL TRIAL: NCT06915480
Title: Reducing Appointment NoShow Through Targeted Pre-appointment Messaging
Brief Title: Reducing Missed Appointments
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00455545
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: All families will be randomized to one of three pre-appointment reminder messages. Additionally, families who are at high risk of experiencing a missed appointment will receive patient navigation services in one of the two departments.
Who Masked: Participant, Care Provider
Masking Description: Families and providers will be fully masked to condition. The investigators will know about condition as they orchestrate the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Standard message, no navigator (Active Comparator): This arm represents the standard operating procedures. It includes basic appointment information and no personal assistance with appointment navigation.
  Interventions: Behavioral: Reminder message and patient navigation
- Standard message with navigator (Experimental): This arm represents the standard pre-appointment reminder message. This arm will include personal assistance with appointment navigation.
  Interventions: Behavioral: Reminder message and patient navigation
- Enhanced message #1, no navigator (Experimental): This arm represents a novel pre-appointment reminder message based on existing scientific literature. This arm will not include personal assistance with appointment navigation.
  Interventions: Behavioral: Reminder message and patient navigation
- Enhanced message #1 with navigator (Experimental): This arm represents a novel pre-appointment reminder message based on existing scientific literature. This arm will include personal assistance with appointment navigation.
  Interventions: Behavioral: Reminder message and patient navigation
- Enhanced message #2, no navigator (Experimental): This arm represents a second novel pre-appointment reminder message based on existing scientific literature. This arm will not include personal assistance with appointment navigation.
  Interventions: Behavioral: Reminder message and patient navigation
- Enhanced message #2 with navigator (Experimental): This arm represents a second novel pre-appointment reminder message based on existing scientific literature. This arm will include personal assistance with appointment navigation.
  Interventions: Behavioral: Reminder message and patient navigation

INTERVENTIONS:
Behavioral: Reminder message and patient navigation — This study will evaluate the combination of pre-appointment messages and patient navigation services.

SUMMARY:
There are four goals of this project: (1) To examine the impact of different appointment reminder messages on appointment attendance; (2) to determine the added benefit of a patient navigator reaching out in advance of appointments to families at elevated risk of missing their appointment, and determine the most common barriers families face in appointment attendance; (3) to evaluate which patients are at highest risk of missing their appointment, and to determine the effectiveness of the intervention trial across different patient risk levels; and (4) to examine if the missing appointment interventions increase the socioeconomic diversity patients.

DETAILED DESCRIPTION:
Aim 1: To test messaging strategies aimed at reducing missed appointments, via a randomized trial, across two different Kennedy Krieger outpatient clinics. Using the reminder system timeline and contact strategy already in effect in these two centers, the investigators will trial alternative language in the reminders (i.e., enhanced message #1 and enhanced message #2) against the current standard of care language. Hypothesis 1: Enhanced messaging will be superior to the standard of care in terms of reducing missed appointments. The investigators do not make a priori hypotheses regarding which enhanced messaging strategy will be optimal, given the exploratory nature.

Aim 2: To determine the added benefit of receiving patient navigation services for families at elevated risk of missing their appointment, and to understand the barriers to child neurodevelopmental evaluation appointments for the purposes of informing future interventions. Throughout the intervention trial, the patient navigator will continuously gather qualitative information on the barriers to appointment attendance faced by families identified to be at elevated risk of missing their evaluation appointment. Understanding these barriers will be critical to the development of future intervention efforts. Hypothesis 2a: Patient navigation services will be superior to enhanced or standard messaging alone in reducing missed appointments. Hypothesis 2b: Most families contacted by the patient navigator will face more than one barrier to attendance, and most barriers will fall into thematic categories that can be used to develop targeted interventions.

Aim 3: To examine the factors related to missed appointments. While the study team has previously identified families that are high-risk for missing their child's appointment, how those family and child-related factors replicate in a novel clinic is unknown. Hypothesis 3: The missing appointment factors will generally reproduce in an independent clinic, Center for Autism (n~3600 yearly diagnostic evaluation appointments), and generally reproduce in the updated data within Center for Neuropsychological and Psychological Assessment (n~6,200 yearly diagnostic evaluation appointments). This will allow the investigators to determine if the intervention is effective particularly for families at elevated risk of missing their appointment (Aim 4).

Aim 4: To examine if the missing appointment interventions increase the socioeconomic diversity of Kennedy Krieger patients. Previous research shows families from less advantaged socioeconomic backgrounds are more likely to miss their appointments. The goal of the intervention is to increase equity among Kennedy Krieger patients, rather than sacrificing equity at the expense of higher show rates (e.g., using punitive procedures). Hypothesis 4: More families at elevated risk of missing their appointments will attend their appointments when receiving the enhanced messages compared to standard messages, and further supported via patient navigation.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled to be seen within the center for autism or the center for neuropsychological and psychological assessment for evaluation appointments will be automatically enrolled in the reminder message portion of the intervention trial.
* Patients who are at elevated risk within the center for neuropsychological and psychological assessment are automatically enrolled in the patient navigator portion of the intervention trial.

Exclusion criteria:

* None for the messaging portion of the study
* For patient navigation, patients >18 years of age will be excluded.

Ages: 1 Month to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient appointment no-show | 6 months
  Proportion of appointments that are neither kept nor cancelled

SECONDARY OUTCOMES:
Patient appointment cancel | 6 months
  Proportion of appointments that are cancelled (>48 hours of appointment date)

CONTACTS AND LOCATIONS:
Overall Officials: luther G kalb, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gornik AE, Northrup RA, Kalb LG, Jacobson LA, Lieb RW, Peterson RK, Wexler D, Ludwig NN, Ng R, Pritchard AE. To confirm your appointment, please press one: Examining demographic and health system interface factors that predict missed appointments in a pediatric outpatient neuropsychology clinic. Clin Neuropsychol. 2024 Feb;38(2):279-301. doi: 10.1080/13854046.2023.2219421. Epub 2023 Jun 8. PMID 37291078
- [Background] Kalb LG, Freedman B, Foster C, Menon D, Landa R, Kishfy L, Law P. Determinants of appointment absenteeism at an outpatient pediatric autism clinic. J Dev Behav Pediatr. 2012 Nov-Dec;33(9):685-97. doi: 10.1097/DBP.0b013e31826c66ef. PMID 23095496
- [Background] Berliner Senderey A, Kornitzer T, Lawrence G, Zysman H, Hallak Y, Ariely D, Balicer R. It's how you say it: Systematic A/B testing of digital messaging cut hospital no-show rates. PLoS One. 2020 Jun 23;15(6):e0234817. doi: 10.1371/journal.pone.0234817. eCollection 2020. PMID 32574181